CLINICAL TRIAL: NCT02148887
Title: Plasticity of Grey and White Matter in Response to Motor Skill Training in Healthy Individuals and Those With Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Foundation Wings For Life (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-2013-0559/PB_2016-00624
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Investigating Spinal Atrophy in Patients With Spinal Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- SCI patients with upper limb impairment - Upper limb training
- SCI patients with lower limb impairment - Lower limb training
- Healthy controls - Upper limb training
- Healthy controls - Lower limb training
- Healthy controls - No intervention

SUMMARY:
We aim to investigate the effect of motor skill training of the upper and lower limbs on the function and structure of the CNS as measured by neuroimaging parameters sensitive to changes in tissue volume and density and the properties of myelin.

DETAILED DESCRIPTION:
Functional recovery following human spinal cord injury (SCI) remains frustratingly limited and the majority of patients are left with severe impairments. While rehabilitative training has been shown to improve clinical outcome following SCI and has a major effect on patients' quality of life, the neuronal mechanisms underpinning neurological and functional recovery are not well understood.

Until recently, degenerative changes in components of the CNS remote to a SCI were thought to occur slowly (over years) and correlate with the degree of disability. Using longitudinal MRI protocols we have shown that these structural changes in fact occur early and progress both at the cord and brain level according to a specific spatial and temporal pattern (Freund et al 2013). It is thought that these trauma-induced structural changes progress retrogradely along central motor nerve fibres of the myelinated corticospinal tract (CST) and this is accompanied over time by shrinkage of corticospinal projecting neuronal bodies. Crucially, patients with less atrophy throughout the CST were those with better clinical recovery at twelve months. Despite this significant recovery advantage in some patients, all participants showed irreversible tissue loss, potentially hindering further recovery. Using the neuroimaging biomarkers established in the previous study cited above, we now aim to assess whether specific and intensive motor learning through tasks for the upper and lower limb might slow or reverse the atrophy seen in the sensorimotor system.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Injury to the spinal cord which leads to any neurological deficits
* able to provide Informed consent

Controls:

- able to provide informed consent

Exclusion Criteria:

* Pregnancy
* MRI incompatible
* Neurologic or physiatric disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with spinal injury
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-02; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
MRI parameters: tensor based morphometry, longitudinal relaxation rate, magnetisation transfer and diffusion index changes in the cervical and cranial corticospinal tract, basal ganglia, motor, premotor and parietal cortex. | MRI scans at weekly intervals (day 0, 7, 14, 28 and 84 after commencement of training)
Raw performance data in the upper and lower limb training task, recorded at each training session. | Training sessions 4x1hour per week for 4 weeks

SECONDARY OUTCOMES:
Overall activity levels as recorded by a worn accelerometer and clinical scoring tests repeated immediately following the first and final training scan sessions (Day 0 and 28) and the 84 day follow-up scan. | Training sessions 4x1hour per week for 4 weeks; clinical assessments at day 0, 28, 84
3D gait analysis will be performed on certain patients and control subjects at the first and final training scan sessions (Day 28) and the 84 day follow-up scan | 3D gait analysis at day 0, 28, 84

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik Balgrist, Zurich, Switzerland